CLINICAL TRIAL: NCT02454842
Title: A Phase 2 Study of TH-4000 (Tarloxotinib) in Patients With EGFR-Mutant, T790M-Negative, Advanced Non-Small Cell Lung Cancer Progressing on an EGFR Tyrosine Kinase Inhibitor
Brief Title: Study for Treatment With TH-4000 (Tarloxotinib) in Epidermal Growth Factor Receptor (EGFR) Mutant, T790M-negative Non-small Cell Lung Cancer (NSCLC) Patients
Acronym: TH-4000
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-601
Record Dates: First submitted 2015-05-04; First posted 2015-05-27 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Non-small Cell Lung Cancer; NSCLC; Non-squamous NSCLC
Keywords: TH-4000; low-oxygen conditions; hypoxia; non-small cell lung cancer; NSCLC; squamous cell carcinoma; Tarloxotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TH-4000 (Tarloxotinib) (Experimental): TH-4000 (Tarloxotinib), 150 mg/m2 will be administered by IV infusion on Days 1, 8, 15, and 22 of each 28-day cycle until progressive disease (PD) or unacceptable toxicity
  Interventions: Drug: TH-4000 (Tarloxotinib)

INTERVENTIONS:
Drug: TH-4000 (Tarloxotinib) — TH-4000 (Tarloxotinib) is a hypoxia-activated prodrug

SUMMARY:
This phase 2 study is designed to evaluate the safety and activity of TH-4000 a hypoxia-activated prodrug, in patients with EGFR-Mutant, T790M-Negative, Advanced NSCLC.

DETAILED DESCRIPTION:
A single arm open label multi-center Phase 2 study in which the pharmacokinetics, safety, tolerability and efficacy of TH-4000 will be assessed in patients with EGFR mutant, T790M negative advanced NSCLC. Patients must have demonstrated progression during EGFR TKI therapy.

Hypoxia PET scans will be obtained in select centers to analyze potential predictors of tumor response.

ELIGIBILITY:
Key Eligibility Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Confirmed recurrent Stage IV NSCLC which progressed while on treatment with EGFR TKI
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Documented evidence of an EGFR mutation known to be associated with an EGFR TKI sensitivity
* No T790M mutation or small cell transformation including an assessment from tumor biopsy obtained while on or subsequent to the most recent EGFR TKI therapy
* Acceptable laboratory results as indicated by protocol
* Acceptable cardiac function as indicated by protocol

Key Exclusion Criteria:

* Receiving medication that prolongs QT interval, with a risk of causing Torsades de Pointes (TdP) unless ECG meets inclusion criteria while on a stable dose of the medication
* Family history of long corrected QT interval (QTc) syndrome
* Symptomatic central nervous system (CNS) lesions
* Radiation therapy within 2 weeks prior to the first dose of study medication
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to the first dose of study medication
* Concurrent active malignancy requiring systemic treatment
* Any other serious uncontrolled medical disorders or psychological conditions that may interfere with study conduct including but not limited to: clinically significant active infection (e.g., tuberculosis, viral hepatitis, human immunodeficiency virus [HIV]), recent (within 6 months) myocardial infarction or unstable angina, congestive heart failure, poorly-controlled hypertension or diabetes, concurrent active malignancy, or psychiatric condition that may interfere with the patient's ability to follow study procedures
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with response rate as evaluated by RECIST criteria | Approximately 12 months

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose
Type of adverse events (AEs) | Up to 30 days after last dose
Severity of adverse events (AEs) | Up to 30 days after last dose
Duration of response (DOR) calculated for all patients achieving an objective response | Approximately 12 months
Progression-free survival (PFS) | Approximately 12 months
Overall Survival (OS) | Approximately 12 months
Time to peak plasma concentration (Tmax) | Cycle 1 Day 1 predose and up to 24 hours post dose
  Time to peak plasma concentration (Tmax), maximum plasma concentration (Cmax), area under concentration-time curve (AUC)
Maximum plasma concentration (Cmax) | Cycle 1 Day 1 predose and up to 24 hours post dose
Area under concentration-time curve (AUC) | Cycle 1 Day 1 predose and up to 24 hours post dose
QTc Interval | Screening, Cycle 1 Day 1, 8, 15 & 22, Day 1 of subsequent cycles

OTHER OUTCOMES:
Hypoxic volume as measured by Positron Emission Tomography (PET) hypoxia imaging | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Liu, Principal Investigator — Georgetown University Hospital Cancer Center
Locations (12):
- United States (11):
  - University of Southern California-Norris, Los Angeles, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of North Carolina Lineberger Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Peter MacCullum, Melbourne, Victoria, Australia